CLINICAL TRIAL: NCT01304186
Title: An Automated, Tailored Information Application for Medication Health Literacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21MH086491 (NIH); R21MH086491 (NIH)
Record Dates: First submitted 2011-02-18; First posted 2011-02-25 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Human Immunodeficiency Virus I Infection
Keywords: Health literacy; HIV; Medication Adherence; IMB Model
MeSH Terms: conditions — Medication Adherence | interventions — Health Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tailored Information (Experimental): Participants in this arm receive the computer-based tailored information application that focuses on improving health literacy related to treatment of HIV infection.
  Interventions: Behavioral: Tailored Information

INTERVENTIONS:
Behavioral: Tailored Information — The intervention comprises a computer-based application designed to provide individually-tailored information to participants in an interactive fashion.
  Other Names: Health literacy

SUMMARY:
The purpose of this study is to evaluate the acceptability and efficacy of a computer-based tailored information application designed to promote health literacy in persons treated for HIV infection. The study hypothesis is that the application will be acceptable and usable for persons treated for HIV infection, and will improve their levels of adherence to antiretroviral medication treatment.

DETAILED DESCRIPTION:
Health literacy is a critically important problem in improving the effectiveness of health care interventions. Patient behaviors essential to the successful treatment of HIV infection, such as high levels of medication adherence, may depend on patients understanding how to take medication, how to solve medication-related problems, and how to cope with medication side effects. An approach that has shown promise in promoting behavior change in HIV+ persons is the Information-Motivation-Behavior Skills (IMB) model. The intervention proposed in this application will implement a health literacy intervention based in part on insights about behavior change drawn from studies of this model. The purpose of the proposed research is to implement this intervention via a computer-based and automated tailored information application. Participants will first complete an automated computer-administered self interview (ACASI) that will assess medication knowledge, disease knowledge likely to be related to motivation, and problem solving skills. Results of this assessment will feed forward to an automated training application that provides individually-tailored training on these topics. This computer-based program will provide training, test understanding, and if necessary reteach and retest. It will also provide printed information for participants to take home to provide ongoing prompts. This study will comprise two phases. In the first, the program will be developed and tested with potential users to assess its usability and detect problems with the wording of materials. In the second phase, participants' health literacy and cognitive status will be evaluated, their adherence to a medication for HIV infection will be assessed using electronic monitoring, and the effects of the program on their adherence will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Currently treated with at least one medication for HIV infection
* No change in target medication anticipated in the next two months
* Able to participate in the study intervention in English

Exclusion Criteria:

* Psychiatric or cognitive disorder of severity sufficient to make the potential participant unable to provide informed consent.
* Not able to participate in the intervention using English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Medication adherence | Four weeks after intervention
  Medication adherence is assessed using electronic monitoring of pill bottle openings via the Medication Event Monitoring System (MEMS) for the month before and the month after participants engage in the study intervention.

SECONDARY OUTCOMES:
Participant self-efficacy | Immediately after completing the intervention (average time: 15 minutes) and four weeks after the intervention
Mood | Immediately after completing the intervention (average time: 15 minutes) and four weeks after the intervention
Elements of the Information, Motivation, and Behavioral Skills Model | Immediately after completing the intervention (average time: 15 minutes) and four weeks after the intervention
  A self-report questionnaire asking participants about their knowledge, motivation, and behavioral skills with respect to HIV infection and its treatment.
Intervention acceptability and usability | Immediately after the intervention (average time: 15 minutes) and four weeks after the intervention
  A questionnaire assessing elements of the Technology Acceptance Model is administered immediately after completing the intervention and four weeks after its completion.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond L Ownby, MD, PhD, Principal Investigator — Nova Southeastern University
Locations (1):
- Ziff Health Clinics, Nova Southeastern University, Fort Lauderdale, Florida, United States

REFERENCES:
- [Result] Ownby RL, Waldrop-Valverde D, Caballero J, Jacobs RJ. Baseline medication adherence and response to an electronically delivered health literacy intervention targeting adherence. Neurobehav HIV Med. 2012 Oct 18;4:113-121. doi: 10.2147/NBHIV.S36549. PMID 23293544
- [Result] Ownby RL, Waldrop-Valverde D, Hardigan P, Caballero J, Jacobs R, Acevedo A. Development and validation of a brief computer-administered HIV-Related Health Literacy Scale (HIV-HL). AIDS Behav. 2013 Feb;17(2):710-8. doi: 10.1007/s10461-012-0301-3. PMID 22961499
- [Derived] Ownby RL, Waldrop-Valverde D, Jacobs RJ, Acevedo A, Caballero J. Cost effectiveness of a computer-delivered intervention to improve HIV medication adherence. BMC Med Inform Decis Mak. 2013 Feb 28;13:29. doi: 10.1186/1472-6947-13-29. PMID 23446180